CLINICAL TRIAL: NCT02125084
Title: Enzalutamide Plus Everolimus in Men With Metastatic Castrate-Resistant Prostate Cancer: A Phase I Study With a Maximum Tolerated Dose Expansion Cohort
Brief Title: Enzalutamide Plus Everolimus in Men With Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 99
Record Dates: First submitted 2014-04-17; First posted 2014-04-29 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
Keywords: Metastatic Prostate Cancer; Castrate-resistant; Enzalutamide; Everolimus
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Everolimus; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus and Enzalutamide (Experimental): Dose Escalation Phase (18 patients): 3-6 patients will be treated at each dose level until the Maximum Tolerated Dose (MTD) is determined.
  * Everolimus: Orally (PO) once daily (dose to be determined;
  * Enzalutamide: 160mg (four 40mg capsules) PO continuous daily dosing.
  Dose Expansion Phase (23 patients): Everolimus and Enzalutamide to be administered using the MTD determined in the dose escalation phase.
  Interventions: Drug: Everolimus; Drug: Enzalutamide

INTERVENTIONS:
Drug: Everolimus
  Other Names: RAD001; Afinitor; Votubia
Drug: Enzalutamide
  Other Names: MDV3100

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a novel combination of agents, enzalutamide and everolimus, for the treatment of patients with metastatic castrate-resistant prostate cancer who have never received prior chemotherapy, or who have previously received docetaxel chemotherapy and have progressive disease.

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase I study with an expansion cohort, in patients with metastatic Castrate-Resistant Prostate Cancer (CRPC) who are chemotherapy-naive or have previously received docetaxel chemotherapy and have progressive disease at the time of study entry. The dose escalation phase of this study will establish the optimum daily dose of everolimus that can be delivered along with a standard daily dose of enzalutamide to patients with metastatic CRPC. Eligible patients must have evaluable (elevated PSA) or measurable disease (per RECIST v1.1). Following completion of the dose escalation phase, an additional cohort of patients will be treated at the maximum tolerated dose (MTD) to give preliminary information regarding the efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

KEY POINTS:

1. Adenocarcinoma of the prostate confirmed histologically.
2. Metastatic disease confirmed by biopsy or imaging studies.
3. Castrate-resistant prostate cancer (i.e., progression of prostate cancer while receiving standard androgen ablation therapy, orchiectomy or luteinizing hormone-releasing hormone [LHRH] antagonist). Castrate levels of serum testosterone must be documented at progression in patients who have not had an orchiectomy.
4. Chemotherapy-naive or previously treated with docetaxel for metastatic prostate cancer.
5. ECOG of 0 to 2.
6. Patients must have progressive metastatic prostate cancer by at least 1 of the following criteria:

   * Progression of measurable lesions defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
   * Bone progression defined by 2 or more new lesions on bone scan.
   * PSA progression is determined by a minimum of two rising PSA levels with an interval of 1 week or greater between each determination. The screening PSA measurement (documenting progression) must be greater than or equal to 2 ng/mL.
7. Adequate hematologic, hepatic and renal function.
8. Adequate coagulation parameters and serum chemistries.
9. Ability to swallow and retain oral medication.
10. Life expectancy of 6 months or greater.
11. Ability to understand the nature of the study and give written informed consent.

Exclusion Criteria:

1. Treatment with more than 2 prior chemotherapy regimens.
2. Previous treatment with enzalutamide or other investigational androgen receptor inhibitors.
3. Previous treatment with PI3K/mTOR inhibitors.
4. Known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or its excipients.
5. Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. For investigational drugs for which 5 half-lives is less than 21 days, a minimum of 10 days between termination of the investigational drug and administration of study drug is required.
6. Most recent chemotherapy ≤21 days from first dose of study treatment and/or patient did not recover from most recent chemotherapy side effects prior to study entry.
7. CNS metastases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of everolimus plus enzalutamide. | 6-8 months
  MTD will be determined by testing increasing doses of everolimus with standard dose enzalutamide in 3-patient dose escalation cohorts. The MTD is defined as the highest dose at which ≤1 of 6 patients experiences a dose-limiting toxicity (DLT) during 1 cycle (28 days) of therapy, assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Prostate-specific antigen (PSA) response rate | every 8 weeks for up to 24 months
  PSA response will be measured by the percent decreased from the reported baseline value. The proportion of patients with documented PSA decreases of 50% and 85% in PSA levels will be reported separately.
Number of patients with serious and non-serious adverse events. | every 4 weeks up to 24 months
  Evaluate the safety of the combination per CTCAE v4.0, every 4 weeks from date of first study treatment until the date of documented progression, up to 24 months.
Pharmacokinetic sampling for everolimus | Cycle 1, Day 1: prior to initial dose and 2hrs post-dose; Cycles 2 and 3, Day 1: prior to initial dose
  Levels of everolimus in blood samples will be collected from patients at selected timepoints prior to dosing during the first 3 cycles of treatment.

SECONDARY OUTCOMES:
Time to PSA progression | every 8 weeks up to 24 months
  Defined as the time from date of first protocol treatment until date of PSA progression. PSA progression is defined as when patient has both a ≥25% increase above the nadir or baseline value and when the absolute increase is ≥2ng/mL.
Overall Response Rate (ORR) | every 8 weeks up to 24 months
  Soft tissue response rate [percentage of complete responders (CR) and partial responders (PR) per RECIST v1.1]
Progression-free survival (PFS) | every 8 weeks up to 24 months
  Restaging will occur every 8 weeks from date of first treatment until date of first progression, or date of death from any cause, whichever comes first - up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Study Chair — SCRI Development Innovations, LLC
Locations (5):
- United States (5):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Center, St. Petersburg, Florida
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee